CLINICAL TRIAL: NCT01860209
Title: Effect of Intermittent Hemodialysis on Sleep Apnea Syndrome and Its Correlation to Nocturnal Rostral Fluid Shift, in End Stage Renal Disease Patients
Brief Title: Effect of Intermittent Hemodialysis on Sleep Apnea Syndrome in End Stage Renal Disease Patients
Acronym: SASinHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Adam Ogna, Centre d'Investigation et Recherche sur le Sommeil (CIRS), Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CIRS-SASinHD
Record Dates: First submitted 2013-05-18; First posted 2013-05-22 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Obstructive Sleep Apnea; Overhydration; End Stage Renal Disease
Keywords: obstructive sleep apnea; overhydration; end stage renal disease; intermittent ambulatory hemodialysis; polysomnography; bioimpedance; leg fluid shift; neck circumference
MeSH Terms: conditions — Sleep Apnea, Obstructive; Water Intoxication; Kidney Failure, Chronic | interventions — Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): the first polysomnography (PSG) is performed before hemodialysis (HD), followed by a post-HD PSG on the subsequent night
  Interventions: Procedure: Hemodialysis
- Group B (Experimental): the first PSG is performed after hemodialysis (HD), followed by a pre-HD PSG, on the subsequent night
  Interventions: Procedure: Hemodialysis

INTERVENTIONS:
Procedure: Hemodialysis — Intermittent ambulatory hemodialysis session, according to the patient usual protocol (defined by the treating nephrologist independently of the study)

SUMMARY:
The purpose of this study is to investigate the effect of decreasing fluid overload by hemodialysis on the severity of obstructive sleep apnea, in patients with end stage chronic kidney disease on intermittent hemodialysis. It aims further to investigate the relationship between overhydration, nocturnal rostral fluid shift and the severity of sleep apnea.

DETAILED DESCRIPTION:
Obstructive sleep disordered breathing is more prevalent in end stage kidney disease patients than in the general population, and may participate to the increased cardiovascular mortality observed in this group of patients. Despite a significant increase in knowledge about the harmful effects of obstructive sleep apnea, the pathophysiological mechanisms are poorly understood. Recent observations suggest a causative relationship between overnight fluid displacement from the legs to the neck soft and the severity of obstructive sleep apnea. This mechanism was demonstrated in otherwise healthy subjects, in heart failure patients, and in patients with venous insufficiency. We thus suspect that this pathophysiologic mechanism could explain the increased prevalence of obstructive sleep apnea in patients with hypervolemia, including chronic renal failure.

The purpose of this trial is to investigate the hypothesis that nocturnal rostral fluid ship is linked to overhydration and participates significantly to the severity of obstructive sleep apnea in patients on hemodialysis. The correction of overhydration by hemodialysis should therefore reduce the amount of nocturnally displaced water and consequently lower the severity of obstructive sleep apnea.

The severity of obstructive sleep apnea is measured by two consecutive attended polysomnographies, performed before and after an ambulatory hemodialysis session with fluid removal, whereas overhydration and leg fluid are evaluated by bioimpedance, performed at the beginning and at the end of each polysomnography. The sequence of the two polysomnographies with respect to hemodialysis is randomized, to minimize the first-night effect.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe obstructive sleep apnea syndrome, with an apnea-hypopnea index (AHI) ≥ 15/h
* age ≥ 18 years
* patient with end stage renal disease on chronic intermittent hemodialysis

Exclusion criteria:

* unstable congestive heart failure
* pace-maker
* active psychiatric disease
* amputation of the lower limbs, proximal to the ankle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Reduction of the obstructive sleep apnea severity | two nights (before and after an ambulatory hemodialysis session)
  Reduction of the obstructive sleep apnea severity, measured by attended polysomnography, after an ambulatory hemodialysis session

SECONDARY OUTCOMES:
Reduction in nocturnal leg fluid volume shift between the legs and the neck | two nights (before and after an ambulatory hemodialysis session)
  Reduction in nocturnal leg fluid volume shift between the legs and the neck, measured by bioimpedance and neck circumference after an ambulatory hemodialysis session
relationship between overhydration, leg fluid volume shift, ankle and neck circumference and the severity of obstructive sleep apnea syndrome | one night
  relationship between overhydration (measured by bioimpedance), leg fluid volume shift, ankle and neck circumference and the severity of obstructive sleep apnea syndrome
severity of the periodic limb movement disorder (PLMD) | two nights (before and after one hemodialysis session)
  severity of the periodic limb movement disorder (PLMD)
severity of central sleep apnea syndrome | two nights (before and after one hemodialysis session)
  severity of central sleep apnea syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Heinzer, MD, Principal Investigator — Centre d'Investigation et Recherche sur le Sommeil (CIRS) - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Switzerland
Locations (1):
- Centre d'Investigation et Recherche sur le Sommeil (CIRS) - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland